CLINICAL TRIAL: NCT05081869
Title: Investigation of the Effect of Online Yoga Based Exercise Program on Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yaren cakmak, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-772.02-E.60605
Record Dates: First submitted 2021-03-26; First posted 2021-10-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Yoga; Telerehabilitation; Exercise; Online
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training; Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Fifty women with primary dysmenorrhea will be divided into two groups as study and control. The working group will be subjected to informative training and an online exercise program of 16 sessions. The control group will only receive information training.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Yoga Based Exercise Program (Experimental): A 50-minute online exercise program consisting of 5 categories will be created. The program will last 8 weeks, twice a week. In the first category, 20-30 seconds of stretching was applied to iliopsoas, hamstring, adductor, tensor fascia lata, piriformis, quadratus lumborum, quadriceps femoris and gastrocnemius muscles. In the second category, stabilization and pelvic mobilization exercises will be applied to the core muscles. Each exercise will be performed in 3 sets of 10 repetitions. In the third category, strengthening exercises will be done for the gluteal muscles, abdominal muscles, erector spine, quadriceps femoris and latissimus dorsi. Each exercise will be performed as 10 repetitions and 3 sets. In the fourth category, 3 sets and 10 repetitions of kegel exercises will be done. minute diaphragmatic breathing will be applied.
  Interventions: Other: Exercise Program; Other: Education Program
- Education Program (Sham Comparator): The informative training was given to both group members individually and online. In the training program; The female reproductive system organs, the structure of the pelvis, the location and functions of the pelvic floor muscles, the definition and physiology of menstruation, the types and risk factors of dysmenorrhea, the definition and symptoms of primary dysmenorrhea, treatment methods for coping with pain in primary dysmenorrhea were mentioned.
  Interventions: Other: Education Program

INTERVENTIONS:
Other: Exercise Program — An online yoga-based exercise program will be applied for 16 sessions in individuals' own environments. The exercise program will consist of stretching, mobilization, stabilization, strengthening and relaxation exercises.
  Arms: Online Yoga Based Exercise Program
Other: Education Program — There will be video training on the subject for both groups.

SUMMARY:
Dysmenorrhea; It is defined as painful menstrual bleeding and is included in the 10th Revision of International Disease Statistics and Related Health Problems published by the World Health Organization in 1992. In women with dysmenorrhea, pain usually begins within 1-2 years after menarche, is intermittent, cramp-like, predominantly in the suprapubic region, and may sometimes be accompanied by various symptoms such as diarrhea, nausea, and vomiting. The incidence of dysmenorrhea can often differ because most women suffering from this problem do not seek any health care services. Symptoms of the menstrual period may negatively affect women in all areas of life by causing various somatic and psychological problems. The state of being absent at least once at school or work due to symptoms of primary dysmenorrhea has been reported by 13-51% of women suffering from this condition. In the treatment of dysmenorrhea, the application of exercise to reduce the level of pain and alleviate the severity of symptoms was started by Mosler in 1914. Mosler demonstrated that exercise pumps blood to the uterus, thereby reducing menstrual pain. In later recent studies, it was found that exercise increases beta-endorphin hormone secretion, which has a natural pain reliever effect in the body; suggested that it reduces stress, pain, and prostaglandin levels. Therefore, the use of exercise as a therapy is thought to improve not only pain and mental health symptoms, but also the quality of life. As of March 11, 2020, since the World Health Organization defined Coronavirus Disease 2019 (COVID-19) as a pandemic. In the current epidemic process, the concept of "social distance" has been emphasized as the most important and basic way of reducing the risk of transmission from close contact, and the importance of choosing telerehabilitation has been emphasized once again. Online application of exercise programs can be defined as telerehabilitation, as the transmission of rehabilitation services over long distances by using electronic information and communication technology. In recent years, it has become one of the popular areas with the development of technology. Due to the limited number of studies on this subject in the literature, our study aimed to investigate the effect of the online yoga-based exercise program on women with primary dysmenorrhea.

DETAILED DESCRIPTION:
This study will be conducted online between March 2021 and May 2021 in their own settings for women with regular menstrual cycles to investigate the impact of online yoga-based exercise programs on women with primary dysmenorrhea. All participants will be given detailed information about the study and a written informed consent form will be signed that they agree to work voluntarily. The GPower program was used to determine the number of people to be included in the study and control groups. When the results of two studies similar to our study were evaluated in the literature review, it was seen that the Effect size d value for the VAS score was distributed between 0.17 and 2.06 and clustered around 1. When the effect size was d = 1, α = 0.05, Power (1-β) = 0.90 (90%) was taken in the GPower package program, and the minimum sample size was determined to be 50, 25 in the study and control groups. They will be randomly divided into two groups of 25 people each, according to the order of application. While an online yoga-based exercise program and an informative training program was applied to the experimental group from two randomly separated groups, only an informative training program will be given to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a nulliparous woman between the ages of 18-35,
* Having a primary dysmenorrhea symptom,
* Having a regular menstrual cycle (28 ± 7 days),
* Menstrual pain Visual Analogue Scale score higher than 4 cm in the last 6 months

Exclusion Criteria:

* Having gastrointestinal, urogynecological, autoimmune, psychiatric, neurological diseases or other chronic pain syndromes,
* To have given birth, Current pregnancy status,
* Using an intrauterine device and having had pelvic surgery,
* Using drugs including oral contraceptives or antidepressants at least 6 months before the study,
* Having an irregular menstrual cycle (those with a menstrual cycle shorter than 21 days or longer than 35 days)
* A pathological history or ultrasonographic result showing secondary dysmenorrhea.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Evaluation | At the baseline
  A personal data questionnaire was used, in which personal information and information about menstrual periods were questioned.
Pain Intensity | Change from Baseline pain intensity at 8 weeks
  Visual Analogue Scale was used to measure the pain intensity. The visual analog scale consists of emotional adjectives that mark the level of pain experienced by the person at that moment with a vertical line on the plane. Participants were asked to rate their menstrual pain levels. Each emotion was evaluated between not experiencing that emotion at all (eg, I'm not nervous = 0) and being fully experienced (eg, I'm extremely nervous = 10).
Life Quality | Change from Baseline life quality at 8 weeks
  Short Form-36 (SF36) questionnaire, evaluates general health and quality of life. The questionnaire has 36 questions and 8 subscales. Limitations in social activities due to physical health-related limitations, physical pain, general health perceptions, vitality, physical or emotional problems and general mental health are questioned. The answers of the questions are scored between 0 (low) and 100 (high). 0 means the lowest level of life and 100 the highest level of quality of life.
Menstrual Attitude | Change from Baseline menstrual attitude at 8 weeks
  The Turkish version of the Menstrual Attitude Scale (MBI) consisting of 5 subscales and a total of 33 items was used to determine the attitudes and behaviors of women during the menstrual period.It was prepared in 1980, based on the view that attitudes about menstruation can be positive as well as negative, and expectations about physiological and emotional symptoms before or during menstruation can be effective in behaviors displayed during this period. Menstruation as a debilitating phenomenon (12 items); Menstruation as a disturbing phenomenon (6 items); Menstruation as a natural phenomenon (5 items); It is a scale consisting of 5 categories and 33 sub-items, including recognizing / anticipating that menstruation will occur (5 items) and denial of the effects of menstruation (7 items). Each item is scored between 1 (strongly disagree) and 5 (totally agree). The high scores obtained from the subscales in the Menstruation Attitude Scale indicate that the attitude towards menstruation
Body Awareness | Change from Baseline body awareness at 8 weeks
  Participants; The Body Awareness Questionnaire, which was developed by Shields et al. In 1989, was used to define body awareness, evaluate the effectiveness of the treatment, and determine its relationship with physical and emotional components. Body Awareness Questionnaire is defined as a tool with psychometric features that fully evaluates the concept of body awareness. It consists of 18 questions in total. Each question is scored between 1 (Not right at all for me) to 7 (Totally true for me). A high score in the questionnaire means high body awareness.
Satisfaction survey | At the end of the 8 weeks
  Three questions about the satisfaction of the online exercise program applied at the end of the study were asked to the participants in the study group. Satisfaction with the treatment and the level of recommending the treatment to other patients were asked to be scored between 0 and 10, and if they had a choice, they were asked whether they would prefer an online or a face-to-face exercise program.
Weight | At the baseline
  kg
Height | At the baseline
  m

CONTACTS AND LOCATIONS:
Overall Officials: Yaren Çakmak, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillen TI, Grbavac SL, Johnston PJ, Straton JA, Keogh JM. Primary dysmenorrhea in young Western Australian women: prevalence, impact, and knowledge of treatment. J Adolesc Health. 1999 Jul;25(1):40-5. doi: 10.1016/s1054-139x(98)00147-5. PMID 10418884
- [Background] Campbell MA, McGrath PJ. Use of medication by adolescents for the management of menstrual discomfort. Arch Pediatr Adolesc Med. 1997 Sep;151(9):905-13. doi: 10.1001/archpedi.1997.02170460043007. PMID 9308868
- [Result] Hasanpour M, Mohammadi MM, Shareinia H. Effects of reflexology on premenstrual syndrome: a systematic review and meta-analysis. Biopsychosoc Med. 2019 Oct 24;13:25. doi: 10.1186/s13030-019-0165-0. eCollection 2019. PMID 31673284
- [Result] Li R, Li B, Kreher DA, Benjamin AR, Gubbels A, Smith SM. Association between dysmenorrhea and chronic pain: a systematic review and meta-analysis of population-based studies. Am J Obstet Gynecol. 2020 Sep;223(3):350-371. doi: 10.1016/j.ajog.2020.03.002. Epub 2020 Mar 7. PMID 32151612
- [Result] Kannan P, Claydon LS, Miller D, Chapple CM. Vigorous exercises in the management of primary dysmenorrhea: a feasibility study. Disabil Rehabil. 2015;37(15):1334-9. doi: 10.3109/09638288.2014.962108. Epub 2014 Sep 22. PMID 25243766
- [Result] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Result] Wosik J, Fudim M, Cameron B, Gellad ZF, Cho A, Phinney D, Curtis S, Roman M, Poon EG, Ferranti J, Katz JN, Tcheng J. Telehealth transformation: COVID-19 and the rise of virtual care. J Am Med Inform Assoc. 2020 Jun 1;27(6):957-962. doi: 10.1093/jamia/ocaa067. PMID 32311034
- [Result] Yonglitthipagon P, Muansiangsai S, Wongkhumngern W, Donpunha W, Chanavirut R, Siritaratiwat W, Mato L, Eungpinichpong W, Janyacharoen T. Effect of yoga on the menstrual pain, physical fitness, and quality of life of young women with primary dysmenorrhea. J Bodyw Mov Ther. 2017 Oct;21(4):840-846. doi: 10.1016/j.jbmt.2017.01.014. Epub 2017 Feb 7. PMID 29037637
- [Result] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- See also: Effects of reflexology on premenstrual syndrome: a systematic review and meta-analysis — http://bpsmedicine.biomedcentral.com/articles/10.1186/s13030-019-0165-0
- See also: Coronavirus disease (COVID-19) pandemic/Vaccines, treatment & tests — http://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Public health matters — http://publichealthmatters.blog.gov.uk/